CLINICAL TRIAL: NCT06696378
Title: Impact of Melatonin Supplementation Plus Exercise Program in Women Who Have Suffered from Breast Cancer in the Province of Soria, Spain
Brief Title: Melatonin Supplementation and Exercise Program in Breast Cancer Women
Acronym: MEXBSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Sanidad de Castilla y León (Other); Ministerio de Ciencia e Innovación, Spain (Other Government); Fundación General Universidad de Valladolid (Other)
Responsible Party: Principal Investigator, Diego Fernández Lázaro, Professor Doctor, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.08.12
Record Dates: First submitted 2024-08-22; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Female Breast Cancer; Older Adults; Exercise Trainning Progrmam
Keywords: Brear Cancer; Melatonin; quality of life; physical performance; health biomarkers; antioxidant capacity; anthropometrics parameters; Exerkins
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Parallel group placebo-controlled randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Double (Investigator, Participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin supplementation group (Experimental): 2 capsules distributed in a single daily oral intake at 9 p.m. or 30 minutes before bedtime, whichever came first, for 10 weeks.
  Interventions: Dietary Supplement: Melatonin 6 mg
- Placebo supplementation group (Placebo Comparator): 2 capsules distributed in a single daily oral intake at 9 p.m. or 30 minutes before bedtime, whichever came first, for 10 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin 6 mg — wo capsules per day; Each capsule includes 3mg Melatonin Nutrifoods® Laboratories, Barcelona, Spain) by the Magistral Formulation Laboratory of a Pharmacy (Soria, Spain), following the rules of the Royal Spanish Pharmacopoeia (Ministry of Health, Government of Spain). Melatonin has a technical data sheet that guarantees its composition and purity (Reference No.: DIE-134).
  Arms: Melatonin supplementation group
Other: Placebo — Two capsules per day; Each capsule includes 100-mg maltodextrin capsules were used as a placebo to match the color and texture of the Melatonin tablets to ensure blinding.
  Arms: Placebo supplementation group

SUMMARY:
Introduction: Breast cancer (BC) remains the leading cause of cancer in women with nearly 1.4 million new cases worldwide annually and 27.000 in Spain. Increasingly effective oncology therapies, however, have numerous adverse effects such as muscle degeneration, fatigue, decreased physical function and aerobic capacity, and deteriorating quality of life. In this sense, physical activity (PA) seems to be an interesting non-pharmacological strategy to alleviate these serious complications and with potential benefits for women with BC. Melatonin (N-acetyl-5 methoxytryptamine) is an indolic compound present with pleiotropic bioactions that regulates the circadian rhythm, antioxidant, anti-inflammatory, immunostimulant, cardioprotective, antidiabetic, antiobesity, neuroprotective, and antiaging actions. Furthermore, in recent years, many studies have described the key role of melatonin in preventing and developing cancer. The general anticarcinogenic mechanisms include epigenetic control, cell proliferation modulation, cell cycle regulation, apoptosis induction, and telomerase inhibition. Melatonin also exerts antiestrogenic activity, which is particularly significant in hormone-dependent tumors, regulating the expression and transactivation of the estrogen receptor, and modulating the enzymes involved in the local synthesis of estrogens. Despite all the mentioned properties, the use of melatonin in daily clinical practice is very limited, and additional studies are needed to better establish the role of this hormone in oncological clinical applications against different types of cancer.

Objective: To analyze the effect of supplementation with 4 g/day of melatonin for 10 weeks on muscle damage (CK and LDH), hormonal responses (estradiol, testosterone, cortisol and testosterone/cortisol ratio), antioxidant capacity (BAP and d-ROMs), Exerkins (Irisin and Sestrin 2), physical performance (handgrip strength, RPE and SPPB), anthropometry (body mass, BMI and fat mass) and WHOQOL-BREF (physical and psychological health, social relationships and environment) in women over 60 years of age who have suffered breast cancer and who follow a physical training program.

Methods: A total of 20 female volunteers between 60 and 73 years old (age: 65.5±4.52 years, BMI: 25.83±2.67 and body fat percentage: 33.73±5.54) who followed a physical activity adapted to their age and abilities are the members. of this study. The volunteers were divided into two groups: placebo (CG; n = 10) and supplemented with 5 g/day of melatonin (GI; n = 10). Differtent test were performed muscle damage (CK, and LDH), hormonal responses (estradiol, testosterone, cortisol, and testosterone/cortisol ratio), antioxidant capacity (BAP and d-ROMs), Exerkins (Irisin and Sestrin 2), physical performance (Hand-grip strength, RPE and SPPB), anthropometrics (Body mass, BMI and fat mass), and WHOQOL-BREF (physical and psychological health, social relationships and environment) were analyzed at the beginning (T1) and at the end of the 10 weeks of intervention (T2).

ELIGIBILITY:
Inclusion Criteria:

* Study participants were women with a history of ductal carcinoma in situ, lobular carcinoma in situ, or stage 1 to 3 breast cancer (5 years or more since diagnosis), not currently receiving chemotherapy or hormone therapy, postmenopausal, and Eastern Cooperative Oncology Group (ECOG) score ≤ 1

Exclusion Criteria:

* women who had exercised regularly for at least 20 minutes once and at least twice a week in the 3 months before the study
* Stage IV breast cancer or systemic recurrences
* Known autoimmune diseases: systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), and multiple sclerosis.
* Severe kidney disease
* Use of adjuvant hormonal therapy, oral estrogen or progesterone replacement therapy, luteinizing hormone-releasing hormone agonists currently or within the past 60 days
* 6-month ≥ post-chemotherapy
* Concomitant use of sleeping pills every night at bedtime
* Concomitant use of black cohosh, flaxseed, or soy in pill or supplement form
* Functional limitation using the Barthel scale (less than 100 = maximum score) and the Lawton-Brody scale (less than 8 = maximum value).
* Uncontrolled hypertension (>180/100 mm Hg).
* Uncontrolled atrial or ventricular arrhythmias, dissecting aortic aneurysm, severe aortic stenosis, acute endocarditis/pericarditis
* Acute thromboembolic disease.
* Moderate/severe chronic obstructive pulmonary disease (COPD) with Bodex index C or D Recent bone fracture (last month).
* Any other circumstance that your doctor considers prevents physical activity.
* Neoadjuvant chemotherapy or radiotherapy
* Concomitant use of beta-blockers
* 6-month ≥ post-radiotherapy
* Concomitant use of postmenopausal hormone replacement therapy
* Use of any type of oral melatonin supplement in the past 30 days
* Acute/chronic heart failure with NYHA (New York Heart Association) score >II
* Uncontrolled orthostatic hypotension
* Recent acute myocardial infarction (3 to 6 months) or unstable angina.
* Acute/chronic respiratory failure.
* Diabetes mellitus with acute decompensation or uncontrolled hypoglycemia
* History of dementia (suspected by the GP environment and diagnosed).
* Shift-work and night-work

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Older women who have suffered from breast cancer
Enrollment: 120 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Irisin | first day of study and after 60 days of supplementation (end of study)
  Exerkin secreted primarily by skeletal muscle in response to exercise
Sestrin-2 | first day of study and after 60 days of supplementation (end of study)
  Exerkin a highly conserved stress-responsive protein, can be triggered by various noxious stimuli, such as hypoxia, DNA damage, oxidative stress, endoplasmic reticulum (ER) stress, and inflammation.

SECONDARY OUTCOMES:
BAP | first day of study and after 60 days of supplementation (end of study)
  biological antioxidant potential (BAP) test to estimate antioxidant capacity by measuring the blood concentration of antioxidants
d-ROMs | first day of study and after 60 days of supplementation (end of study)
  diacron reactive oxygen metabolites (d-ROMs) pro-oxidant state of a biological sample, measures hydroperoxides
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | first day of study and after 60 days of supplementation (end of study)
  a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment
Creatine kinase (CK) | first day of study and after 60 days of supplementation (end of study)
  CK is an enzyme expressed by various tissues and cell types; markers of muscle damage
Lactate dehydrogenase (LDH) | first day of study and after 60 days of supplementation (end of study)
  LDH is a catalytic enzyme found in many tissues of the body;markers of muscle damage
Cortisol | first day of study and after 60 days of supplementation (end of study)
  catabolic hormone released in response to stress
Testosterone | first day of study and after 60 days of supplementation (end of study)
  anabolic hormone
Estradiol | first day of study and after 60 days of supplementation (end of study)
  female sex hormone of the estrogen group.
BMI | first day of study and after 60 days of supplementation (end of study)
  Body Mass Index (BMI) anthropometric parameter which is the relationship between a person's body mass and their height
Fat Mass | first day of study and after 60 days of supplementation (end of study)
  Anthropometric parameter fat mass allows the estimation of overweight or obesity in humans
Short Physical Performance Battery (SPPB) | first day of study and after 60 days of supplementation (end of study)
  Test evaluates three aspects of mobility measures balance, the second gait speed, and the third leg strength
Hand-grip strength | first day of study and after 60 days of supplementation (end of study)
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles
RPE-Borg 10 | first day of study and after 60 days of supplementation (end of study)
  RPE stands for Rating of Perceived Exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, University of Valladolid Soria Campus, Soria, Soria, Spain

REFERENCES:
- [Derived] Celorrio San Miguel AM, Cacharro LM, Santamaria G, Garrosa M, Celorrio San Miguel M, Roche E, Garrosa E, Fernandez-Lazaro D. Adjuvant melatonin therapy during exercise prescription in breast cancer survivors on physical and anthropometric parameters, quality of life, and hormonal response. A randomized controlled trial. Front Sports Act Living. 2025 Jun 23;7:1594733. doi: 10.3389/fspor.2025.1594733. eCollection 2025. PMID 40625889